CLINICAL TRIAL: NCT05989919
Title: Nasal Anatomical and Pathological Variants in Patients With Antrochoanal Polyps
Status: Completed | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Maisara Mohamed, assistant lecturer of otorhinolaryngology, Minia University
Other Study IDs: 538-2022
Record Dates: First submitted 2023-08-05; First posted 2023-08-14 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Antrochoanal Polyp

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: patients with antrochoanal polyps
  Interventions: Other: CT scan for nose and paranasal sinuses
- control group: patients with unilateral sinonasal disease other than antrochoanal polyps
  Interventions: Other: CT scan for nose and paranasal sinuses

INTERVENTIONS:
Other: CT scan for nose and paranasal sinuses — CT scan for nose and paranasal sinuses

SUMMARY:
The goal of this observational study is to learn about anatomical and pathological variants in patients with antrochoanal polyps trying to find a key to its pathogenesis Participants will have nasal endoscopic examination and CT nose and paranasal sinuses.

we will compare patients with antrochoanal polyps and other patients with unilateral sinonasal disease regarding anatomical and pathological variants.

DETAILED DESCRIPTION:
This study was conducted at Otolaryngology department, Minia University Hospital, Minia, Egypt. The study was approved by the Institutional Review Board at Minia University.

The study participants were recruited from patients complaining from unilateral sinonasal disease attending outpatient clinic.

we selected 40 patients with ACPs who had the following inclusion criteria: 1-radiologically diagnosed based on CT nose and PNS. 2-histopathologically diagnosed as ACP. The radiological diagnosis is based on seeing low attenuated soft tissue mass filling the maxillary antrum and extending through the middle meatus into the nasal cavity and directs towards the post nasal opening. We excluded: 1- patients with history of maxillofacial trauma. 2- patients who had previous nasal surgery.

To be more objective, a control group of 40 patients who had unilateral sinonasal disease other than ACP was formed.

We assessed multislice computed tomography (CT) nose and paranasal sinus images by Toshiba aquilion CT scanner. Axial and coronal 250mm cuts were obtained.

Both study and control groups were compared regarding anatomical and pathological variations in the nose. These variants include: deviated nasal septum, concha bullosa, paradoxical middle turbinate and uncinate process insertion (to lamina papyrecea or roof of ethmoid or middle turbinate). We also compare between them according to presence of retention cyst in CT in contralateral side In the cases with deviated nasal septum, the septal deviation was seen if it is towards the side of the lesion or towards the opposite side according to its convexity.

We also evaluate the sclerosis on thickening of the bony wall of the para nasal sinus as an indication of chronic inflammation.

SPSS 24.0 program was used for statistical analysis. Averages and standard deviations were calculated. The Mann-Whitney and Chi square tests were used for comparisons between the groups. The Pearson correlation tests was used to evaluate correlations. Statistical significance was set at ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. radiologically diagnosed based on CT nose and PNS.
2. histopathologically diagnosed as ACP.

Exclusion Criteria:

1. patients with history of maxillofacial trauma.
2. patients who had previous nasal surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study participants were recruited from patients complaining from unilateral sinonasal disease attending our outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
presence of anatomical and pathological variants in CT scan and endoscopic examination | 6 months
  Both study and control groups were compared regarding anatomical and pathological variations in the nose. These variants include: deviated nasal septum, concha bullosa, paradoxical middle turbinate and uncinate process insertion (to lamina papyrecea or roof of ethmoid or middle turbinate). We also compare between them according to presence of retention cyst in CT in contralateral side In the cases with deviated nasal septum, the septal deviation was seen if it is towards the side of the lesion or towards the opposite side according to its convexity.
  We also evaluate the sclerosis on thickening of the bony wall of the para nasal sinus as an indication of chronic inflammation.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided